CLINICAL TRIAL: NCT04937049
Title: Effectiveness and Usability of a Web Tool for the Self-management of Women's Health Needs During Pregnancy, Childbirth and the Puerperium: EMAeHealth
Brief Title: EMAehealth Web Tool for Pregnancy and Puerperium: Effectiveness
Acronym: EMAeHealthEF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Biobizkaia Health Research Institute (Other Government)
Collaborators: Carlos III Health Institute (Other Government); Basque Health Service (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: EMAeHealth effectiveness
Record Dates: First submitted 2021-06-11; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Pregnant Women; Postpartum Period
Keywords: women; pregnancy; puerperium; eHealth; Antenatal Education; Health needs; Web tool

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMAeHealth digital tool (Experimental): This team has designed a digital tool called EMAeHealth involving healthcare professionals. It is organized into 4 areas: 1) an Information area, 2) a Communication area, 3) a Health Self-management area, 4) a Clinical data area, The tool is conceived as a complement that can reinforce maternal health education with resources that facilitate its accessibility, and rapid remote response, which will also improve its results. It will be incorporated into the Osakidetza-Basque Health Service corporate Website.
  Interventions: Other: EMAeHealth digital tool
- No EMAeHealth digital tool (No Intervention): Usual care. This group, like experimental group, receives the usual care, which includes traditional maternal education, but does not receive the EMAeHealth intervention

INTERVENTIONS:
Other: EMAeHealth digital tool — eHealth intervention to support Maternal Education
  Arms: EMAeHealth digital tool

SUMMARY:
The research team has designed, and will test, a web tool to support traditional Maternal Education (EM). This tool is organized into 4 areas: 1) Information área; 2) Communication área (with peers and with professionals) 3) Self-management health area(instruments to check or reflect on their own health needs, as well as decision algorithms to detect the time of delivery and postpartum alarm symptoms); 4) Clinical data área (the woman can have her clinical data, include it and share it with other professionals) The objective of the study is to evaluate the clinical effectiveness of the EMAeHealth tool and also its implementation in the real world (its usability and acceptability, by women and professionals).

DETAILED DESCRIPTION:
The usefulness of Maternal Education, as it is currently being developed, is being questioned due to the obvious changes that have arisen in access to information by mothers and fathers, and due to the changes that have occurred in childbirth care and in the attitude towards the process of motherhood and fatherhood. There is no doubt, however, about the need to advise, care for and accompany couples in this stage of physical, family and social change. To respond to these new needs, the evidence indicates that a digital format may be the most appropriate. So, the research team has designed, and intends to test, a web tool, which is organized into 4 areas: 1) Information area: which will have information based on evidence, permanently updated by health services professionals ; 2) Communication area: allows women to contact other women in similar circumstances, through forums or conversations, or consult with professionals 3) Self-management health area : who have valid and reliable self-assessment instruments to check their own health needs, as well as decision algorithms to detect the time of delivery and postpartum alarm symptoms; 4) Clinical data area: in which the woman can collect clinical data, include the most recent and share it with other professionals if she so wishes. The first area is open access, but not the other three, which require a password. The objective is to evaluate the clinical effectiveness of the EMAeHealth tool, and also its implementation in the real world (its usability and acceptability, by women and professionals). Methods: The research team propose a hybrid implementation-effectiveness design, which allows us to evaluate aspects related to the context while evaluating the clinical efficacy of the tool. Discussion: A tool like the one described is of interest to women, to professionals and also to the health system. Note- Clinical Trials submision correspond to clinical effectiveness part of the study. Usability and acceptability is not included because it use qualitative methods.

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman
* week 8-10 of gestation
* to speak and understand Spanish language

Exclusion Criteria:

• not meeting any of the inclusion criteria

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1080 (Estimated)
Dates: Start 2022-01-10 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is change from baseline in Health-related quality of life, measured with the Spanish version of the Short Form 36 Health Survey | 9 months.Measurements: at weeks 8th(baseline) and 37th of pregnancy, and at weeks 1th, 6th, and 16th postpartum
  The Spanish version of the SF-36 questionnaire assess the health-related quality of life.It´s made up of 8 domains, of which 4 are oriented towards physical aspects and another 4 towards mental aspects of health-related quality of life. Two summaries are made of this physical and mental component, which explain between 80 and 85% of the variance. The scores of the questionnaire are transformed on a scale from 0 to 100 points; the higher the score, the better the perception of health-related quality of life. A difference of 5 points in the domain score, or between 2 and 3 points in the summary score is considered clinically relevant. Vilagut G, 2005. doi:10.1157/13074369

SECONDARY OUTCOMES:
Change from baseline in Self-efficacy for labor and childbirth, measured with the Spanish version of Lowe's Childbirth Self-Efficacy Inventory scales. | 29 weeks. Measurements alt 8th(baseline) and 37th of pregnancy.
  The Childbirth Self-Efficacy Inventory (CBSEI) was developed by Nancy K Lowe in USA.The inventory is a self-report instrument that includes 62- items. It is divided into four subscales measuring both outcome expectancies, i.e. what behavior they think would be useful during labour as well as self-efficacy expectancies, i.e. how they think they will be able to conduct themselves during labour. The instrument measures these two dimensions of the self-efficacy construct, during both the first and the second stage of the labour process. The responses are distributed by a 15-item scale for the outcome expectancy scales and a 16-item scale for the self-efficacy expectancy scales. The response rates for all four scales range from 1 to 10; higher scores indicate a higher degree of childbirth self-efficacy. (Cunqueiro MJ, et al Childbirth Self-Efficacy Inventory: psychometric testing of the Spanish version. J Adv Nurs. 2009;65(12):2710-2718. doi:10.1111/j.1365-2648.2009.05161.x)
Change from baseline in Self-efficacy for breasfeeding, measured with The Spanish version of the Breastfeeding Self-Efficacy Scale-Short Form | 16 weeks. Measurements: at 1th(baseline), 6th and 16 weeks of portpartum period.
  The Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) was developed to measure a mother's confidence in her ability to breastfeed her new infant. The BSES-SF is a 14-item, unidimensional, self-report instrument developed to measure a mother's confidence in her ability to breastfeed. All items are presented positively and anchored with a 5-point Likert-type scale where 1 indicates not at all confident and 5 indicates always confident. Higher scores indicate higher levels of breastfeeding self-efficacy. The translated Spanish version of BSES-SF scale can be considered a valid and reliable measure of maternal breastfeeding self-efficacy in Spain. (Oliver-Roig A et al, Dennis The Spanish version of the Breastfeeding Self-Efficacy Scale-Short Form: reliability and validity assessment. Int J Nurs Stud. 2012;49(2):169-173. doi:10.1016/j.ijnurstu.2011.08.005)

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Artieta, PHD, Principal Investigator — Osakidetza- Basque HS

IPD SHARING:
Plan to Share IPD: Yes
The protocol and the research results will be published.
  Access to the data is feasible by requesting permission from the main researcher, Isabel Artieta
  The protocol and the research results will be published.
  Access to the data is feasible by requesting permission from the main researcher, Isabel Artieta
  The protocol and the research results will be published. Access to data, ICF, etc. are available by requesting it from the main researcher, Isabel Artieta (MARIAISABEL.ARTIETAPINEDO@osakidetza.eus )
Supporting Information: Study Protocol, CSR
Time Frame: 2023-2024
Access Criteria: The protocol and the research results will be published. Access to data, ICF, etc. are available by requesting it from the main researcher, Isabel Artieta (MARIAISABEL.ARTIETAPINEDO@osakidetza.eus )

REFERENCES:
- [Result] Vilagut G, Ferrer M, Rajmil L, Rebollo P, Permanyer-Miralda G, Quintana JM, Santed R, Valderas JM, Ribera A, Domingo-Salvany A, Alonso J. [The Spanish version of the Short Form 36 Health Survey: a decade of experience and new developments]. Gac Sanit. 2005 Mar-Apr;19(2):135-50. doi: 10.1157/13074369. Spanish. PMID 15860162
- [Result] Cunqueiro MJ, Comeche MI, Docampo D. Childbirth Self-Efficacy Inventory: psychometric testing of the Spanish version. J Adv Nurs. 2009 Dec;65(12):2710-8. doi: 10.1111/j.1365-2648.2009.05161.x. PMID 19941552
- [Result] Oliver-Roig A, d'Anglade-Gonzalez ML, Garcia-Garcia B, Silva-Tubio JR, Richart-Martinez M, Dennis CL. The Spanish version of the Breastfeeding Self-Efficacy Scale-Short Form: reliability and validity assessment. Int J Nurs Stud. 2012 Feb;49(2):169-73. doi: 10.1016/j.ijnurstu.2011.08.005. Epub 2011 Sep 17. PMID 21930270
- [Derived] Espinosa Cifuentes M, Artieta-Pinedo I, Paz-Pascual C, Bully-Garay P, Garcia-Alvarez A; ema-Q Group. EMAeHealth, a digital tool for the self-management of women's health needs during pregnancy, childbirth and the puerperium: protocol for a hybrid effectiveness-implementation study. BMJ Open. 2022 Sep 1;12(9):e055031. doi: 10.1136/bmjopen-2021-055031. PMID 36575817